CLINICAL TRIAL: NCT05172700
Title: Expanded Access Program for Pirtobrutinib for Previously Treated B-Cell Cancers
Brief Title: Expanded Access Program for Pirtobrutinib for Participants With B-Cell Cancer
Status: Approved for marketing | Type: Expanded Access
Sponsor: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Other Study IDs: 17712; J2N-OX-Y001 (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-12-15; First posted 2021-12-29 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Lymphocytic, Small; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia; Ritcher's Transformation, Syndrome
Keywords: BTKi; BTK Inhibitor; Bruton's tyrosine kinase inhibitor; Hematologic Disease; B-cell receptor
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia; Syndrome; Hematologic Diseases | interventions — pirtobrutinib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Pirtobrutinib — Administered orally.
  Other Names: LY3527727; LOXO-305

SUMMARY:
This is an expanded access program for eligible participants with a previously treated B-cell cancer who are ineligible for an ongoing pirtobrutinib clinical trial.

The treating physician/investigator contacts Lilly when, based on their medical opinion, a patient meets the criteria for inclusion in the expanded access program.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with:

  * CLL or SLL and have received treatment with the following five classes of therapy: Chemotherapy, anti-cluster of differentiation (anti-cd) 20 antibody, covalent Bruton's tyrosine kinase (BTK) inhibitor, B-cell lymphoma-2 (BCL-2) inhibitor, and phosphatidylinositol 3-kinase (PI3K) inhibitor
  * MCL that has been previously treated with a covalent BTK inhibitor
  * Richter's Transformation (RT) with previous Richter's directed-therapy
  * Waldenstrom macroglobulinemia (WM), previously treated with chemotherapy, anti-CD20 antibody and a covalent BTK inhibitor
* Are not eligible for an ongoing pirtobrutinib clinical trial

Exclusion Criteria:

* Inadequate organ function
* Significant cardiovascular disease
* History of allogenic or autologous stem cell transplant (SCT) or chimeric antigen receptor modified Tcell (CAR-T) therapy within 60 days
* Tested positive for human immunodeficiency syndrome (HIV) or known active hepatitis B or C virus or cytomegalovirus (CMV) infection
* Active, uncontrolled autoimmune cytopenia
* Clinically significant active malabsorption syndrome
* Participants requiring therapeutic anticoagulation with warfarin or another vitamin K antagonist

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Contact Lilly at 1-800-LillyRx (1-800-545-5979), Study Director — Eli Lilly and Company